CLINICAL TRIAL: NCT04370834
Title: Tocilizumab in Hospitalized Cancer Patients With Coronavirus 2019 (SARS-CoV-2) and Severe Complications of Coronavirus Disease 19 (COVID-19)
Brief Title: Tocilizumab for Patients With Cancer and COVID-19 Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - Randomized data no longer support continuation
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCI-2020-02987; NCI-2020-02987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); TRC-10446 (Other: National Cancer Institute); TRC-10446 (Other: CTEP)
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Results first posted 2021-06-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm; Pneumonia; Pneumonitis; Severe Acute Respiratory Distress Syndrome; Symptomatic COVID-19 Infection Laboratory-Confirmed
MeSH Terms: conditions — Hematologic Neoplasms; Pneumonia; Respiratory Distress Syndrome | interventions — tocilizumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Other (tocilizumab) (Experimental): Patients receive tocilizumab IV over 60 minutes. A second dose may be given if there is sustained or recurrent fever, no decrease or not more than a 1-category improvement on the 7-category ordinal scale (only stabilization or partial improvement following first dose), or a >= 1-category worsening on the 7-category ordinal scale from nadir.
  Interventions: Biological: Tocilizumab

INTERVENTIONS:
Biological: Tocilizumab — Given IV
  Other Names: Actemra; Immunoglobulin G1, Anti-(Human Interleukin 6 Receptor) (Human-Mouse Monoclonal MRA Heavy Chain), Disulfide with Human-Mouse Monoclonal MRA Kappa-Chain, Dimer; MRA; R-1569; RoActemra

SUMMARY:
This phase II expanded access trial will study how well tocilizumab works in reducing the serious symptoms including pneumonitis (severe acute respiratory distress) in patients with cancer and COVID-19. COVID-19 is caused by the SARS-CoV-2 virus. COVID-19 can be associated with an inflammatory response by the immune system which may also cause symptoms of COVID-19 to worsen. This inflammation may be called "cytokine storm," which can cause widespread problems in the body. Tocilizumab is a medicine designed to block the action of a protein called interleukin-6 (IL-6) that is involved with the immune system and is known to be a key factor for problems with excessive inflammation. Tocilizumab is effective in treating "cytokine storm" from a type of cancer immunotherapy and may be effective in reducing the inflammatory response and "cytokine storm" seen in severe COVID-19 disease. Treating the inflammation may help to reduce symptoms, improve the ability to breathe without a breathing machine (ventilator), and prevent patients from having more complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To enhance access to tocilizumab for patients who cannot participate in the randomized COVACTA trial with specific emphasis on patients with cancer, especially those who belong to high-risk and minority populations and children.

II. To provide observations on clinical outcomes associated with tocilizumab administration in cancer patients with severe acute respiratory syndrome (SARS) coronavirus 2 (COVID-19) disease.

SECONDARY OBJECTIVE:

I. To estimate the proportion of patients whose level of institutional care does not further escalate following administration of tocilizumab.

EXPLORATORY OBJECTIVES:

I. To estimate the number of days intensive care unit (ICU) patients spent in the ICU.

II. To evaluate the mortality rate of patients:

IIa. 30-day and 60-day mortality in patients in the ICU.

IIb. Evaluate the 14-, 30- and 60-day mortality rate following infusion of tocilizumab.

III. To evaluate overall survival.

IV. To describe the proportion of patients progressing to ventilator support after tocilizumab therapy.

V. Evaluate the clinical course following administration of tocilizumab.

Va. To evaluate the development of additional infections.

Vb. To evaluate the side effects following tocilizumab.

Vc. To evaluate impact on inflammatory markers.

VI. Evaluate the duration of time:

VIa. To removal from mechanical ventilator support.

VIb. To step-down of institutional care requirements.

VIc. To discharge from the ICU to lower level.

VId. To hospital discharge.

VIe. To resolution of clinical symptoms.

VIf. To time of defervescence.

VIg. To normalization of disease-related laboratory abnormalities.

VII. Exploratory biologic correlates.

VIIa. To evaluate cytokine levels pre and post-tocilizumab, specifically evaluating IL-6.

VIIb. To evaluate SARS-coronavirus (CoV)-2 viral loads pre and post-tocilizumab.

VIIc. To determine the pharmacokinetics of tocilizumab in order to facilitate exposure-response analysis.

VIId. To correlate clinical outcomes with changes in cytokine levels and SARS-CoV-2 viral loads.

OUTLINE:

Patients receive tocilizumab intravenously (IV) over 60 minutes. A second dose may be given if there is sustained or recurrent fever, no decrease or not more than a 1-category improvement on the 7-category ordinal scale (only stabilization or partial improvement following first dose), or a >= 1-category worsening on the 7-category ordinal scale from nadir.

After completion of study treatment, patients are followed up for at least 60 days, and, when possible, up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have an active cancer diagnosis or have completed therapy within 12 months of initiation of protocol specified therapy. This includes:

  * Subjects with a new cancer diagnosis who have not yet initiated cancer therapy
  * Subjects on active or have recently completed cancer-directed therapy including chemotherapy, radiation therapy, immunotherapy or hormonal therapy amongst others

    * Myelosuppressive chemotherapy for patients in remission (e.g., adjuvant chemotherapy for breast cancer, acute myeloid leukemia [AML] consolidation) is prohibited until clinical recovery (1 or 2 on the 7-category ordinal scale)
  * Subjects on any investigational therapy for their underlying cancer, investigational COVID-19 anti-viral agents, or convalescent serum aimed at treating COVID-19 disease are eligible. Investigators are reminded to check whether the other investigational study(s) the patient is participating on specifically exclude tocilizumab and to adjudicate best clinical management decision for the specific patient
  * Subjects who have undergone hematopoietic stem cell transplant within the past 12 months, or are continued on graft versus host disease (GVHD) therapy, are also eligible
* COVID-19 Diagnosis: Patients hospitalized with COVID-19 pneumonia confirmed by:

  * Radiographic findings concerning for COVID-19 pneumonia AND
  * Confirmatory SARS-CoV-2 positive result using any testing assay, or (with or without a confirmatory test) with suspicion of COVID-19 disease owing to belonging to a high-risk demographic group or living and/or working in high-risk settings or with known exposure AND
  * Oxygen saturation (SpO2) on room air =< 93% or PaO2/FiO2 < 300 mmHg
* Age >= 2 years
* Patients must have adequate organ function as assessed by the treating investigator to administer tocilizumab
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 10 x institutional upper limit of normal
* Patients with low blood counts attributable to cancer therapy or underlying malignancy are eligible
* Patients may be on other therapies for COVID-19 including investigational and not limited to corticosteroids, azithromycin, chloroquine, hydroxychloroquine

  * For patients already enrolled on other investigational studies for COVID-19, study investigators should verify that co-enrollment on this study is permissible as per the eligibility of the other study
* Human immunodeficiency virus (HIV)-infected patients are eligible for this trial unless they have opportunistic complications of acquired immunodeficiency syndrome (AIDS) other than the cancer they have
* For patients with evidence of chronic hepatitis B virus (HBV) infection, should be on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection should be on treatment if indicated
* The effects of tocilizumab on the developing human fetus are unknown

  * Pregnancy: Based on animal data, may cause fetal harm. Tocilizumab may be given if in the physician's judgment the patient's life is threatened without potential effective therapy

    * Women of childbearing potential must agree to use birth control or remain abstinent for the duration of the study and for at least 28 days following the last dose of tocilizumab. Pregnancy tests should be done based on the discretion of the patient and physician.
    * Nursing mothers: Discontinue drug or nursing taking into consideration importance of drug to mother
    * Men must agree to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agree to refrain from donating sperm, for the duration of the study and for at least 28 days following the last dose of tocilizumab
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Prior or concurrent utilization of IL-6 specific targeting strategies for treatment of COVID-19 that showed no benefit after maximum dosing; (patients who have only received 1 prior dose and there was evidence of potential benefit may be eligible)

  * This includes siltuximab, tocilizumab, and sarilumab
* Known hypersensitivity or history of severe allergic reaction to tocilizumab or other monoclonal antibodies
* Any serious medical condition or active uncontrolled infections (besides COVID-19) that, in the investigator's judgement, preclude the subject's safe participation in the study

  * Examples: Active tuberculosis (TB) infection
* Active diverticulitis because of severe flairs in disease leading risk of bowel perforation
* Patients in whom, in the opinion of the treating physician, progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments, will be excluded from the study
* Patients receiving or planning to receive any investigational agents other than tocilizumab are ineligible for this study, with the following exceptions:

  * Investigational agents directed at a patient's underlying cancer are allowed.
  * Investigational SARS-CoV-2 anti-viral agents
  * Convalescent serum directed at COVID-19 disease

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard F Little, Principal Investigator — National Cancer Institute (NCI)
Locations (5):
- United States (5):
  - National Cancer Institute, Rockville, Maryland
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Valley Medical Center, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Other (Tocilizumab)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Other (Tocilizumab)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Cohort [Count of Participants; unit: Participants]
  Cohort A1 | 1
  Cohort A2 | 0
  Cohort B1 | 0
  Cohort B2 | 0
Cancer type [Count of Participants; unit: Participants]
  Hematologic | 1
  Solid tumor | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Point Reduction in Score on 7-category Clinical Status Ordinal Scale
Description: 7-category Clinical Status Ordinal Scale:
  1. Discharge
  2. Non-ICU, hospital ward, No O2
  3. Non-ICU, hospital ward, on O2
  4. ICU or non-ICU, requires non-invasive ventilatory support or high flow O2
  5. ICU requires mechanical or imminent ventilation/intubation
  6. ICU requires ECMO and additional O2 support and organ support, e.g. vasopressors, renal replacement therapy
  7. Death
Time Frame: Day 14 after tocilizumab administration
Population: No patients were accrued to Cohorts A2, B1, or B2.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A1: Clinical Status Ordinal Scale 3-4, Not on mechanical ventilation at time of registration and no immediate plan for intubation, At least 30 kg
- Cohort A2: Clinical Status Ordinal Scale 3-4, Not on mechanical ventilation at time of registration and no immediate plan for intubation, Less than 30 kg
- Cohort B1: Clinical Status Ordinal Scale 5-6, On mechanical ventilation at time of enrollment or imminent intubation indicated, At least 30 kg
- Cohort B2: Clinical Status Ordinal Scale 5-6, On mechanical ventilation at time of enrollment or imminent intubation indicated, Less than 30 kg
Arm/Group | Cohort A1 | Cohort A2 | Cohort B1 | Cohort B2
Number analyzed (Participants) | 1 | 0 | 0 | 0
Participants | 1 |  |  |

ADVERSE EVENTS:
Time Frame: 30 days after tocilizumab administration
Description: One patient was enrolled to this trial. This patient enrolled to Cohort A1.
Arm/Group | Cohort A1 | Cohort A2 | Cohort B1 | Cohort B2
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=1) | Cohort A2 (N=0) | Cohort B1 (N=0) | Cohort B2 (N=0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 (N=1) | Cohort A2 (N=0) | Cohort B1 (N=0) | Cohort B2 (N=0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination as randomized data did not support continuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04370834/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04370834/ICF_001.pdf